CLINICAL TRIAL: NCT05569525
Title: Effects of Non-surgical Periodontal Therapy on the Glycemic Variability of Periodontal Patients Affected by Type I Diabetes. a Randomized Clinical Trial.
Brief Title: Type I Diabetes and Non-surgical Periodontal Treatment
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florence (Other)
Responsible Party: Principal Investigator, Dr. Francesco Cairo, Prof., University of Florence
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIODO
Record Dates: First submitted 2022-10-03; First posted 2022-10-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Type 1 Diabetes; Periodontitis; Periodontal Diseases; Diabetes; Diabetes Mellitus; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Periodontitis; Periodontal Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Patients receiving non-surgical periodontal treatment within 1 week from enrollment.
  Interventions: Procedure: Non-surgical periodontal therapy
- Control (Active Comparator): Patients receiving non-surgical periodontal treatment 6 months after the enrollment.
  Interventions: Procedure: Non-surgical periodontal therapy

INTERVENTIONS:
Procedure: Non-surgical periodontal therapy — Non-surgical periodontal therapy according to the full-mouth debridement protocol.

SUMMARY:
Current evidence suggests a bidirectional association between periodontitis and diabetes. Periodontal therapy improves short term HbA1c levels and is safe to perform. Most studies are focused on type 2 Diabetes. Literature about the correlation between periodontitis and type 1 diabetes is scarce, since no randomized clinical trials have been performed.

The objective of the present clinical investigation is to evaluate the effects of nonsurgical treatment of periodontal disease on glycemic variability in patients with type 1 diabetes (T1DM). The hypothesis is that nonsurgical periodontal therapy affects glycemic variability in terms of time spent in hyperglycemia.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 1 diabetes
* Patients under treatment in the department of Diabetology of AOU Careggi having a microinfusor for continuous subcutaneous insulin infusion (CSII) and a Flash Glucose Monitoring (FGM) device
* Diagnosis of periodontitis (all stages and grades)

Exclusion Criteria:

* Contraindications for non-surgical periodontal therapy
* Pregnancy
* History of other systemic disease (cancer, HIV, bone metabolic dysease, Head and Neck Radiotherapy, Immunosuppressive/modulating therapy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-06 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) | 6 months after the non-surgical periodontal treatment
  Glycated hemoglobin (HbA1c) to evaluate glycemic variability measured as a percentage (%).

SECONDARY OUTCOMES:
Standard Deviation (SD) of glycaemia | 6 months after the non-surgical periodontal treatment
  Standard Deviation: the spread of glucose readings around the average (mg/dl)
Glucose coefficient of variability (CV) | 6 months after the non-surgical periodontal treatment
  CV is a calculation: dividing the SD by the mean glucose and multiplying by 100 to get a percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Università degli Studi di Firenze, Florence, FI, Italy

IPD SHARING:
Plan to Share IPD: No